CLINICAL TRIAL: NCT05592028
Title: Bilateral Transcranial Magnetic Resonance-guided Focused Ultrasound Pallidothalamic Tractotomy for Patients With X-linked Dystonia-parkinsonism
Brief Title: High Intensity Focused Ultrasound for X-linked Dystonia-parkinsonism
Status: Available | Type: Expanded Access
Sponsor: University of the Philippines Manila - Philippine General Hospital (Other)
Responsible Party: Principal Investigator, Roland Dominic G. Jamora, Associate Professor, University of the Philippines Manila - Philippine General Hospital
Other Study IDs: DoN-001
Record Dates: First submitted 2022-08-21; First posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-08

CONDITIONS: X-Linked Dystonia Parkinsonism
Keywords: High intensity focused ultrasound; pallidothalamic tractotomy; transcranial MR-guided focused ultrasound
MeSH Terms: conditions — Dystonia 3, Torsion, X-Linked

STUDY DESIGN:
Expanded Access Types: Individual, Intermediate, Treatment

INTERVENTIONS:
Device: transcranial magnetic resonance-guided focused ultrasound pallidothalamic tractotomy — XDP patients will receive unilateral or bilateral transcranial magnetic resonance-guided focused ultrasound pallidothalamic tractotomy.

SUMMARY:
X-linked dystonia-parkinsonism (XDP) is a rare, X-linked, adult-onset, and progressive movement disorder seen almost exclusively in men from Panay Island in the Philippines. The disease is associated with mutations involving the DYT3/TAF1 gene, and all the cases described so far have been linked to Filipino ancestry. Although XDP is very rare globally, the prevalence is 5.74 per 100,000 individuals in Panay Island and 0.31 per 100,000 in the Philippines as a whole. Majority of patients (95%) were males, and the mean age of onset was 39 years. The mean duration of illness was 16 years, and the mean age of death was 55.6 years.

DETAILED DESCRIPTION:
To determine the outcomes of MRgFUS pallidothalamic tractotomy on adult XDP patients at the Philippine General Hospital.

This is a prospective study that aims to determine the outcomes of MRgFUS pallidothalamic tractotomy (both unilateral and bilateral) on adult XDP patients at the Philippine General Hospital.

No sample size will be determined a priori. The study will be conducted over a period of five years, and all eligible patients may be invited to join the study during this period.

The procedure will be performed inside the MRI suite, using a 1.5 Tesla MRI system (GE Optima MR450, USA) and the ExAblate Neuro device (InSightec, Haifa, Israel) to deliver the focused ultrasound. The patient's head will be shaved and immobilized using a stereotactic frame under local anesthesia. An elastic diaphragm will be attached to the patient's head and connected to the ultrasound transducer,8 and the patient will be positioned inside the bore of the MRI. A reference MRI scan will be performed to position the transducer to the target, after which the MRI images (T1-weighted axial and T2-weighted axial/coronal MRI at 1 mm slices) will be fused to the preoperative CT scan for the skull-correction algorithm.8 Stereotactic treatment planning will then be performed to target the pallidothalamic tract. It is usually located at the midcommisural line (0 to 1.0 mm posterior) in the anterior-posterior direction, 8-10 mm lateral to the intercommisural line in the mediolateral direction, 0-1.5 mm inferior to the intercommisural line in the dorsoventral direction, and 6.5-7.5 mm to the thalamo-ventricular border.7 The lesion will be made 3 mm lateral to the mamillo-thalamic tract and superior and medial to the medial subthalamic nucleus.9,11,12 Once the target is set, a series of low-power sonications producing temperatures between 40-45oC and lasting 10-20 seconds will be performed.8 Clinical assessment for tremor suppression and treatment side effects will be made after each sonication,8 and definitive non-reversible thermal ablation will be performed only at the setting wherein the patient experiences tremor reduction or suppression with no adverse effects.9 The final sonication temperature usually ranges between 55-63oC.8 After the treatment, the stereotactic frame will be removed and the patient will be monitored in the hospital overnight.

The patients will be assessed within 24 hours of treatment then asked to follow up with the movement disorder neurologist (RDJ) at 2 weeks, 3 months, 6 months, 9 months, and 12 months post-treatment through a clinic visit. Video recording will be taken on initial visit and at each follow up visit. Another blinded assessor will score the videos of the patients. The outcome will be assessed using the XDP-Movement Disorder Society of the Philippines (XDP-MDSP) Scale at each visit, and comparing it to the pre-treatment baseline, as well as using the XDP Clinical and Functional Staging. The pre- and post-treatment BFMDRS and UPDRS scores will also be obtained.

For bilateral MRgFUS tractotomy, the contralateral lesion will be done at least 6 months after the first procedure, provided that there are no serious adverse effects from the first PTT lesioning.

Demographic, clinical, treatment-related, and outcome data of all study patients will be collected prospectively by the investigators throughout the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and above
* have been diagnosed with XDP and confirmed by genetic testing
* have a skull density ratio (SDR) of >/= 0.35 on CT scan
* have psychiatric and medical clearance
* have passed the neurocognitive test
* have undergone MRgFUS pallidothalamic tractomy, either unilateral or bilateral,

Exclusion Criteria:

* patients aged less than 18 years old
* patients who have movement disorders other than XDP
* patients with abnormal neuroimaging findings that would preclude MRgFUS lesioning
* Skull SDR < 0.35
* patients with medical contraindications
* patients who did not fulfill the inclusion criteria

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Roland Dominic G Jamora, MD, PhD, Principal Investigator — Department of Neurosciences, University of the Philippines Manila
Locations (1):
- Philippine General Hospital, Manila, Philippines

REFERENCES:
- [Derived] Jamora RDG, Khu KJO, Sy MCC, Pascual JSG, Legaspi GD, Aguilar JA. Transcranial magnetic resonance-guided focused ultrasound pallidothalamic tractotomy for patients with X-linked dystonia-parkinsonism: a study protocol. BMC Neurol. 2023 Aug 18;23(1):306. doi: 10.1186/s12883-023-03344-x. PMID 37596524